CLINICAL TRIAL: NCT06159699
Title: New Challenges for the Population on the Path to Achieving Active Longevity: an Online Survey of Respondents Using Telecommunication Technologies
Brief Title: Telecommunication Technology-based Online Survey
Status: Recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Nina D. Anfinogenova, Principal Investigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Other Study IDs: CRI-248
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Risk Factors; Polypharmacy; Drug Interactions; Self Medication; COVID-19
Keywords: Polypharmacy; Potential Drug-Drug Interactions; Self Medication; COVID-19; Medical Imaging; Environmental Risk Factors; Protracted Low-Dose-Rate Radiation Exposure
MeSH Terms: conditions — COVID-19 | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-structured population: The respondent will represent the non-structured population of the Russian Federation invited to participate in the study using the SMS-Target tool provided by OOO T2 Mobile Company.
  Interventions: Other: Online Survey; Diagnostic Test: Genetic Testing

INTERVENTIONS:
Other: Online Survey — The participants of the study undergo the online survey at www.zdorov.tpu.ru and www.zdorov.expert.
  Other Names: Telecommunication-Based Survey
Diagnostic Test: Genetic Testing — Genetic testing will be performed in subgroup of survey respondents willing to participate in the study of polymorphisms of genes involved in drug metabolism or affecting biological effects of medications including CYP2D6, ACE, UGT1A1, CYP2C9, and CYP2C19.
  Other Names: Genetic Polymorphisms of Drug-Metabolizing Enzymes

SUMMARY:
The aim of this study is to identify and assess new health-associated risk factors, including clinical-pharmacological risk factors. The cohort is built using telecommunication approaches. The associations between clinical-pharmacological, social, demographic, behavioral, and environmental characteristics will be assessed. The continuous depersonalized online survey is performed using the original informational resources in the form of specially designed web-site aimed at identification and assessment of population-based pharmacotherapy patterns including characteristics of self-medication, biologically active food supplement intake, polypharmacy, and adverse drug-drug interactions in the people residing in the ecological conditions of various regions of the country. The invitations to participate in the online survey are sent via the SMS messages using the SMS-Target tool provided by OOO T2 Mobile Company. The survey is performed online at www.zdorov.tpu.ru and www.zdorov.expert both specifically designed for questionnaire publication and data accumulation.

DETAILED DESCRIPTION:
Polypharmacy-associated serious drug-drug interactions and adverse drug reactions may increase the risk of morbidity and mortality in the population, especially in cardiovascular patients. Insufficient patient compliance to treatment and potential self-medication overlap with behavioral, psychosocial, demographic, and environmental conditions and pose new challenges for the population striving to achieve active longevity. These issues have been especially relevant during and after the COVID-19 pandemic. The aim of this study is to identify and assess new health-associated risk factors, including clinical-pharmacological risk factors. Telecommunication approaches are used for the formation of study cohort. The associations between clinical-pharmacological, social, demographic, behavioral, and environmental characteristics of study cohort will be assessed. The continuous depersonalized online survey is performed using the original informational resource in the form of specially designed web-site aimed at identification and assessment of population-based pharmacotherapy patterns including characteristics of self-medication, biologically active food supplement intake, polypharmacy, and adverse drug-drug interactions in the people residing in the ecological conditions of various regions of the country. The acquired data may lay a foundation for the development decision support system for control of previously unrecognized or poorly recognized risk factors. The study will enroll as least 2000 respondents aged 18 years and older. The invitations to participate in the online survey are sent via the SMS messages using the SMS-Target tool provided by OOO T2 Mobile Company. The survey is performed online at www.zdorov.tpu.ru and www.zdorov.expert both specifically designed for questionnaire publication and data accumulation. Both websites have built-in functionality for downloading survey results in tabular format (.xls, .csv). All the respondents are required to sign the informed consent form electronically according to local legislation and international standards of ethical research. Considering that no physical medical examinations or interventions are involved in the study, and all data undergo complete depersonalization, participation in this study does not pose any risks for respondents. Financial support for the study is provided by the Russian Science Foundation (project No. 22-15-00313). Respondents will not be covered by insurance due to the non-interventional nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years and older
* signing the informed concent form online
* completion of the entire questionnaire

Exclusion Criteria:

* age under 18 years
* refuse to sign the informed concent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nonstructured population aged 18 years and older willing to complete the entire questionnaire and signing the informed concent form.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious drug-drug interactions (percent) | Five years
  Incidence of serious drug-drug interactions (DDIs) is assessed as a percentage (%) of completed survey questionnaires associated with serious DDIs relative to the size of respondent population.
Median number of serious drug-drug interactions (n) | Five years
  Median number of serious drug-drug interactions is assessed per one completed survey questionnaire containing information on pharmacotherapy.

SECONDARY OUTCOMES:
Incidence of polypharmacy (percent) | Five years
  Polypharmacy refers to using five or more medications. Incidence of polypharmacy is assessed as a percentage (%) of completed survey questionnaires reporting polypharmacy relative to the size of respondent population.
Incidence of MRI administration (percent) | Two years
  Incidence of magnetic resonance tomography (MRI) administration is assessed as a percentage (%) of completed survey questionnaires where respondents report the fact of undergoing MRI procedure for the past two years relative to the size of respondent population.
Incidence of CT administration (percent) | Two years
  Incidence of computed tomography (CT) administration is assessed as a percentage (%) of completed survey questionnaires where respondents report the fact of undergoing CT procedure for the past two years relative to the size of respondent population.
Incidence of diagnostic ultrasound administration (percent) | Two years
  Incidence of diagnostic ultrasound administration is assessed as a percentage (%) of completed survey questionnaires where respondents report the fact of undergoing ultrasonography procedure for the past two years relative to the size of respondent population.
Incidence of diagnostic X-ray administration (percent) | Two years
  Incidence of diagnostic X-ray administration is assessed as a percentage (%) of completed survey questionnaires where respondents report the fact of undergoing X-ray for the past two years relative to the size of respondent population.
Incidence of scintigraphy administration (percent) | Two years
  Incidence of scintigraphy administration is assessed as a percentage (%) of completed survey questionnaires where respondents report the fact of undergoing scintigraphy for the past two years relative to the size of respondent population.
Incidence of chest fluoroscopy administration (percent) | Two years
  Incidence of chest fluoroscopy administration is assessed as a percentage (%) of completed survey questionnaires where respondents report the fact of undergoing chest fluoroscopy for the past two years relative to the size of respondent population.
Clinically significant CYP2D6 gene polymorphisms | Two months
  Clinically significant CYP2D6 gene polymorphisms will be identified by diagnostic sequencing using EDTA whole blood.
Clinically significant ACE gene polymorphisms | Two months
  Clinically significant ACE gene polymorphisms will be identified by real-time PCR with melting curve detection using EDTA whole blood.
Clinically significant UGT1A1 gene polymorphisms | Two months
  Clinically significant UGT1A1 gene polymorphisms will be identified by real-time PCR with melting curve detection using EDTA whole blood.
Clinically significant CYP2C9 gene polymorphisms | Two months
  Clinically significant CYP2C9 gene polymorphisms will be identified by real-time PCR with melting curve detection using EDTA whole blood.
Clinically significant CYP2C19 gene polymorphisms | Two months
  Clinically significant CYP2C19 gene polymorphisms will be identified by real-time PCR with melting curve detection using EDTA whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Nina D Anfinogenova, PhD, Principal Investigator — Tomsk NRMC
Locations (1):
- Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia